CLINICAL TRIAL: NCT04436640
Title: A Multicenter, Open-Label Extension Study to Asses the Long-Term Safety, Tolerability, and Efficacy of Bimekizumab in the Treatment of Study Participants With Active Axial Spondyloarthritis, Ankylosing Spondylitis, and Nonradiographic Axial Spondyloarthritis
Brief Title: A Study to Evaluate the Long-term Safety, Tolerability and Efficacy of Bimekizumab in Subjects With Active Axial Spondyloarthritis Including Ankylosing Spondylitis and Nonradiographic Axial Spondyloarthritis
Acronym: BE MOVING
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS0014; 2019-004163-47 (EudraCT Number); 2023-506527-28 (Registry Identifier: EU Clinical Trials); U1111-1304-6865 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Axial Spondyloarthritis; Ankylosing Spondylitis; r-axSpa; Nr-axSpa
Keywords: AxSpa; Radiographic; Non-radiographic; AS; Bimekizumab; Axial spondyloarthritis; Ankylosing spondylitis
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bimekizumab (Experimental): Subjects will receive bimekizumab throughout the Treatment Period.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at prespecified time-points.
  Other Names: BKZ; UCB4940

SUMMARY:
The purpose of the study is to demonstrate the long-term safety, tolerability and efficacy of bimekizumab in patients with active axial spondyloarthritis (axSpA, also known as radiographic axSpa (r-axSpA)) including ankylosing spondylitis (AS) and nonradiographic axial spondyloarthritis (nr-axSpa).

ELIGIBILITY:
Inclusion Criteria:

* Study participant is considered reliable and capable of adhering to the protocol (eg, able to understand and complete questionnaires), visit schedule, and medication intake according to the judgement of the Investigator
* In the opinion of the Investigator, the study participant is expected to benefit from participation in this extension study
* Study participant completed AS0010 (NCT03928704) or AS0011 (NCT03928743)

Exclusion Criteria:

* Female study participants who plan to become pregnant during the study or within 20 weeks following final dose of Investigational Medicinal Product (IMP). Male study participants who are planning a partner pregnancy during the study or within 20 weeks following the final dose
* Study participants who meet any withdrawal criteria in AS0010 or AS0011. For any study participant with an ongoing serious adverse event (SAE), or a history of serious infections (including hospitalizations) in the feeder study, the Medical Monitor must be consulted prior to the study participant's entry into AS0014
* Study participant has a positive or indeterminate interferon gamma release assay (IGRA) in AS0010 or AS0011, unless appropriately evaluated and treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events (TEAEs) during the study | From Baseline (Day 1) until Safety Follow-Up (up to Week 180)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Percentage of participants with serious adverse events (SAEs) during the study | From Baseline (Day 1) until Safety Follow-Up (up to Week 180)
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalisation or prolongation of existing hospitalisation
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment with parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardise the patients, or may require medical or surgical intervention to prevent any of the above
Percentage of participants with with treatment-emergent adverse Events (TEAEs) leading to withdrawal from the study | From Baseline (Day 1) until Safety Follow-Up (up to Week 180)
  Treatment-emergent adverse events (TEAEs) are any untoward medical incidence in a subject during administered study treatment, whether or not these events are related to study treatment.

SECONDARY OUTCOMES:
Assessment of SpondyloArthritis International Society 40% response criteria (ASAS40) response at Week 28 | Week 28
  ASAS40 will be calculated relative to Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743). The Assessment of SpondyloArthritis International Society (ASAS) criteria for 40% improvement are defined as relative improvements of at least 40%, and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains and no worsening at all in the remaining domain.
  The domains are:
  * Patient's Global Assessment of Disease Activity (PGADA)
  * Pain assessment (the total spinal pain, NRS score)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))-
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) question 5 and 6 concerning morning stiffness intensity and duration)
Assessment of SpondyloArthritis International Society 40% response criteria (ASAS40) response at Week 52 | Week 52
  ASAS40 will be calculated relative to Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743). The Assessment of SpondyloArthritis International Society (ASAS) criteria for 40% improvement are defined as relative improvements of at least 40%, and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains and no worsening at all in the remaining domain.
  The domains are:
  * Patient's Global Assessment of Disease Activity (PGADA)
  * Pain assessment (the total spinal pain, NRS score)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI))
Assessment of SpondyloArthritis International Society 40% response criteria (ASAS40) response at Week 112 | Week 112
  ASAS40 will be calculated relative to Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743). The Assessment of SpondyloArthritis International Society (ASAS) criteria for 40% improvement are defined as relative improvements of at least 40%, and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 domains and no worsening at all in the remaining domain.
  The domains are:
  * Patient's Global Assessment of Disease Activity (PGADA)
  * Pain assessment (the total spinal pain, NRS score)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI))
Assessment of SpondyloArthritis International Society 20% response criteria (ASAS20) response at Week 28 | Week 28
  ASAS20 will be calculated relative to Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743). The Assessment of SpondyloArthritis International Society (ASAS) criteria for 20% improvement are defined as relative improvements of at least 20%, and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 following domains and absence of deterioration in the potential remaining domain.
  The domains are:
  * Patient's Global Assessment of Disease Activity (PGADA)
  * Pain assessment (the total spinal pain, NRS score)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI))
Assessment of SpondyloArthritis International Society 20% response criteria (ASAS20) response at Week 52 | Week 52
  ASAS20 will be calculated relative to Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743). The Assessment of SpondyloArthritis International Society (ASAS) criteria for 20% improvement are defined as relative improvements of at least 20%, and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 following domains and absence of deterioration in the potential remaining domain.
  The domains are:
  * Patient's Global Assessment of Disease Activity (PGADA)
  * Pain assessment (the total spinal pain, NRS score)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI))
Assessment of SpondyloArthritis International Society 20% response criteria (ASAS20) response at Week 112 | Week 112
  ASAS20 will be calculated relative to Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743). The Assessment of SpondyloArthritis International Society (ASAS) criteria for 20% improvement are defined as relative improvements of at least 20%, and absolute improvement of at least 1 unit on a 0 to 10 Numeric Rating Scale (NRS) in at least 3 of the 4 following domains and absence of deterioration in the potential remaining domain.
  The domains are:
  * Patient's Global Assessment of Disease Activity (PGADA)
  * Pain assessment (the total spinal pain, NRS score)
  * Function (represented by Bath Ankylosing Spondylitis Functional Index (BASFI))
  * Inflammation (the mean of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI))
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 28 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 28
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is a validated self-reported instrument, which consists of six 10-unit horizontal Numeric Rating Scales (NRS) to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI score ranges from 0 to 10, with lower scores indicating lower disease activity.
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 52 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 52
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is a validated self-reported instrument, which consists of six 10-unit horizontal Numeric Rating Scales (NRS) to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI score ranges from 0 to 10, with lower scores indicating lower disease activity.
Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 112 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 112
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is a validated self-reported instrument, which consists of six 10-unit horizontal Numeric Rating Scales (NRS) to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI score ranges from 0 to 10, with lower scores indicating lower disease activity.
Assessment of SpondyloArthritis International Society partial remission (ASAS-PR) at Week 28 | Week 28
  The Assessment of SpondyloArthritis International Society partial remission (ASAS-PR) is defined as a score of <=2 units on a 0 to 10 unit scale in all 4 domains listed for ASAS40 domains.
Assessment of SpondyloArthritis International Society partial remission (ASAS-PR) at Week 52 | Week 52
  The Assessment of SpondyloArthritis International Society partial remission (ASAS-PR) is defined as a score of <=2 units on a 0 to 10 unit scale in all 4 domains listed for ASAS domains.
Assessment of SpondyloArthritis International Society partial remission (ASAS-PR) at Week 112 | Week 112
  The Assessment of SpondyloArthritis International Society partial remission (ASAS-PR) is defined as a score of <=2 units on a 0 to 10 unit scale in all 4 domains listed for ASAS domains.
Assessment of Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) at Week 28 | Week 28
  The ASDAS-C-Reactive Protein (ASDAS-CRP) consists of a number of assessments which are scored by the study participant and physician and multiplied by a proven formula as shown below:
  0.121 x Total back pain (represented by the BASDAI Question 2 result) 0.058 x Duration of morning stiffness (represented by the BASDAI Question 6 result) 0.110 x PGADA 0.073 x Peripheral pain/swelling (represented by the BASDAI Question 3 result) 0.579 x (natural logarithm of the hs-CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue are all assessed on a numerical scale (0 to 10 units). The sum of these weighted components gives the ASDAS-CRP.
Assessment of Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) at Week 52 | Week 52
  The ASDAS-C-Reactive Protein (ASDAS-CRP) consists of a number of assessments which are scored by the study participant and physician and multiplied by a proven formula as shown below:
  0.121 x Total back pain (represented by the BASDAI Question 2 result) 0.058 x Duration of morning stiffness (represented by the BASDAI Question 6 result) 0.110 x PGADA 0.073 x Peripheral pain/swelling (represented by the BASDAI Question 3 result) 0.579 x (natural logarithm of the hs-CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue are all assessed on a numerical scale (0 to 10 units). The sum of these weighted components gives the ASDAS-CRP.
Assessment of Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) at Week 112 | Week 112
  The ASDAS-C-Reactive Protein (ASDAS-CRP) consists of a number of assessments which are scored by the study participant and physician and multiplied by a proven formula as shown below:
  0.121 x Total back pain (represented by the BASDAI Question 2 result) 0.058 x Duration of morning stiffness (represented by the BASDAI Question 6 result) 0.110 x PGADA 0.073 x Peripheral pain/swelling (represented by the BASDAI Question 3 result) 0.579 x (natural logarithm of the hs-CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue are all assessed on a numerical scale (0 to 10 units). The sum of these weighted components gives the ASDAS-CRP.+ 1)
Assessment of SpondyloArthritis International Society (ASAS) 5/6 response at Week 28 | Week 28
  The Assessment of SpondyloArthritis International Society (ASAS) 5/6 response is defined as achieving at least 20% improvement in 5 of 6 domains, including the 4 domains defined for ASAS40 domains as well as spinal mobility (lateral spinal flexion) and high sensitivity C-reactive Protein (hs-CRP).
Assessment of SpondyloArthritis International Society (ASAS) 5/6 response at Week 52 | Week 52
  The Assessment of SpondyloArthritis International Society (ASAS) 5/6 response is defined as achieving at least 20% improvement in 5 of 6 domains, including the 4 domains defined for ASAS domains as well as spinal mobility (lateral spinal flexion) and high sensitivity C-reactive Protein (hs-CRP).
Assessment of SpondyloArthritis International Society (ASAS) 5/6 response at Week 112 | Week 112
  The Assessment of SpondyloArthritis International Society (ASAS) 5/6 response is defined as achieving at least 20% improvement in 5 of 6 domains, including the 4 domains defined for ASAS domains as well as spinal mobility (lateral spinal flexion) and high sensitivity C-reactive Protein (hs-CRP).
Change from Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 28 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 28
  The Bath Ankylosing Spondylitis Functional Index (BASFI) assesses physical function in comprising 10 items relating to activities during the past week. Each item ranges from 0 ('Easy') to 10 ('Impossible'). The BASFI is the mean of the 10 scores such that the total score ranges from 0 to 10, with lower scores indicating better physical function. A negative value in BASFI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Change from Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 52 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 52
  The Bath Ankylosing Spondylitis Functional Index (BASFI) assesses physical function in comprising 10 items relating to activities during the past week. Each item ranges from 0 ('Easy') to 10 ('Impossible'). The BASFI is the mean of the 10 scores such that the total score ranges from 0 to 10, with lower scores indicating better physical function. A negative value in BASFI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Change from Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 112 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 112
  The Bath Ankylosing Spondylitis Functional Index (BASFI) assesses physical function in comprising 10 items relating to activities during the past week. Each item ranges from 0 ('Easy') to 10 ('Impossible'). The BASFI is the mean of the 10 scores such that the total score ranges from 0 to 10, with lower scores indicating better physical function. A negative value in BASFI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Change from Baseline in Nocturnal Spinal Pain Numeric Rating Scale (NRS) at Week 28 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 28
  Nocturnal spinal pain experienced by ankylosing spondylitis (AS) subjects is measured by one question: pain in the spine at night due to AS?. When responding, the subject is to consider the average amount of pain in the preceding week. It is assessed on a numerical scale (0 to 10 units). A lower score indicates less pain and an improvement of the outcome.
Change from Baseline in nocturnal Spinal Pain Numeric Rating Scale (NRS) at Week 52 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 52
  Nocturnal spinal pain experienced by ankylosing spondylitis (AS) subjects is measured by one question: pain in the spine at night due to AS?. When responding, the subject is to consider the average amount of pain in the preceding week. It is assessed on a numerical scale (0 to 10 units). A lower score indicates less pain and an improvement of the outcome.
Change from Baseline in Nocturnal Spinal Pain Numeric Rating Scale (NRS) at Week 112 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 112
  Nocturnal spinal pain experienced by ankylosing spondylitis (AS) subjects is measured by one question: pain in the spine at night due to AS?. When responding, the subject is to consider the average amount of pain in the preceding week. It is assessed on a numerical scale (0 to 10 units). A lower score indicates less pain and an improvement of the outcome.
Change from Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) at Week 28 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 28
  The Ankylosing Spondylitis Quality of Life (ASQoL), a validated disease-specific 18-item questionnaire, has been developed specifically for measuring health-related quality of life (HRQoL) in subjects with ankylosing spondylitis (AS) and has shown to be responsive in axial spondyloarthritis (axSpA). The ASQoL score ranges from 0 to 18 with a higher score indicating worse HRQoL.
Change from Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) at Week 52 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 52
  The Ankylosing Spondylitis Quality of Life (ASQoL), a validated disease-specific 18-item questionnaire, has been developed specifically for measuring health-related quality of life (HRQoL) in subjects with ankylosing spondylitis (AS) and has shown to be responsive in axial spondyloarthritis (axSpA). The ASQoL score ranges from 0 to 18 with a higher score indicating worse HRQoL.
Change from Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) at Week 112 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 112
  The Ankylosing Spondylitis Quality of Life (ASQoL), a validated disease-specific 18-item questionnaire, has been developed specifically for measuring health-related quality of life (HRQoL) in subjects with ankylosing spondylitis (AS) and has shown to be responsive in axial spondyloarthritis (axSpA). The ASQoL score ranges from 0 to 18 with a higher score indicating worse HRQoL.
Change from Baseline in the Short Form 36-Item Health Survey (SF-36) physical component summary (PCS) at Week 28 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 28
  There are 8 Short-Form 36-item Health Survey (SF-36) domain scores. In addition to domain scores, the Physical Component Summary (PCS) scores are calculated from the 8 domains. Each of the 8 domain scores and the component summary scores ranging from 0 to 100, with higher scores indicating better health status. A larger positive value in change from Baseline indicates an improvement.
Change from Baseline in the Short Form 36-Item Health Survey (SF-36) physical component summary (PCS) at Week 52 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 52
  There are 8 Short-Form 36-item Health Survey (SF-36) domain scores. In addition to domain scores, the Physical Component Summary (PCS) scores are calculated from the 8 domains. Each of the 8 domain scores and the component summary scores ranging from 0 to 100, with higher scores indicating better health status. A larger positive value in change from Baseline indicates an improvement.
Change from Baseline in Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) at Week 28 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 28
  The Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) characterizes the spinal mobility of subjects with axial Spondyloarthritis (SpA) and Ankylosing Spondylitis (AS). It is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 is calculated for each item based on the measurement. The mean of the 5 scores provides the BASMI score. The higher the BASMI score the more severe the patient's limitation of movement due to their axial SpA. A negative value in BASMI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Change from Baseline in Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) at Week 52 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 52
  The Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) characterizes the spinal mobility of subjects with axial Spondyloarthritis (SpA) and Ankylosing Spondylitis (AS). It is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 is calculated for each item based on the measurement. The mean of the sum of the 5 scores provides the BASMI score. The higher the BASMI score the more severe the patient's limitation of movement due to their axial SpA. A negative value in BASMI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Change from Baseline in Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) at Week 112 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 112
  The Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) characterizes the spinal mobility of subjects with axial Spondyloarthritis (SpA) and Ankylosing Spondylitis (AS). It is a disease-specific measure consisting of 5 clinical measures to reflect subject axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 is calculated for each item based on the measurement. The mean of the sum of the 5 scores provides the BASMI score. The higher the BASMI score the more severe the patient's limitation of movement due to their axial SpA. A negative value in BASMI change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Change from Baseline in the Maastricht Ankylosing Spondylitis Enthesitis (MASES) Index at Week 28 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 28
  The Maastricht Ankylosing Spondylitis Enthesitis (MASES) is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process) each scored as 0 or 1 and then summed for a possible score of 0 to 13. A higher score indicates worsening.
Change from Baseline in the Maastricht Ankylosing Spondylitis Enthesitis (MASES) Index at Week 52 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 52
  The Maastricht Ankylosing Spondylitis Enthesitis (MASES) is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process) each scored as 0 or 1 and then summed for a possible score of 0 to 13. A higher score indicates worsening.
Change from Baseline in the Maastricht Ankylosing Spondylitis Enthesitis (MASES) Index at Week 112 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 112
  The Maastricht Ankylosing Spondylitis Enthesitis (MASES) is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process) each scored as 0 or 1 and then summed for a possible score of 0 to 13. A higher score indicates worsening.
Change from Baseline in the Short Form 36-Item Health Survey (SF-36) physical component summary (PCS) at Week 112 | From Baseline of AS0010 (NCT03928704) or AS0011 (NCT03928743) to Week 112
  There are 8 Short-Form 36-item Health Survey (SF-36) domain scores. In addition to domain scores, the Physical Component Summary (PCS) scores are calculated from the 8 domains. Each of the 8 domain scores and the component summary scores ranging from 0 to 100, with higher scores indicating better health status. A larger positive value in change from Baseline indicates an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (75):
- United States (10):
  - As0014 50062, Glendale, Arizona
  - As0014 50052, Phoenix, Arizona
  - As0014 50060, Upland, California
  - As0014 50059, Ormond Beach, Florida
  - As0014 50056, Sarasota, Florida
  - As0014 50015, Hagerstown, Maryland
  - As0014 50016, St Louis, Missouri
  - As0014 50055, Portland, Oregon
  - As0014 50020, Duncansville, Pennsylvania
  - As0014 50057, Dallas, Texas
- Belgium (3):
  - As0014 40004, Brussels
  - As0014 40003, Genk
  - As0014 40001, Ghent
- Bulgaria (4):
  - As0014 40006, Plovdiv
  - As0014 40007, Plovdiv
  - As0014 40005, Sofia
  - As0014 40008, Sofia
- China (9):
  - As0014 20040, Beijing
  - As0014 20021, Chengdu
  - As0014 20019, Guangzhou
  - As0014 20034, Hefei
  - As0014 20024, Nanjing
  - As0014 20018, Shanghai
  - As0014 20020, Shanghai
  - As0014 20026, Shanghai
  - As0014 20025, Wenzhou
- Czechia (8):
  - As0014 40011, Brno
  - As0014 40009, Pardubice
  - As0014 40013, Prague
  - As0014 40014, Prague
  - As0014 40015, Prague
  - As0014 40016, Prague
  - As0014 40010, Uherské Hradiště
  - As0014 40012, Zlín
- France (2):
  - As0014 40018, Boulogne-Billancourt
  - As0014 40022, Limoges
- Germany (6):
  - As0014 40025, Berlin
  - As0014 40029, Hamburg
  - As0014 40024, Hanover
  - As0014 40027, Herne
  - As0014 40078, Leipzig
  - As0014 40026, Ratingen
- Hungary (3):
  - As0014 40032, Debrecen
  - As0014 40031, Szeged
  - As0014 40033, Székesfehérvár
- Japan (11):
  - As0014 20035, Bunkyō City
  - As0014 20030, Chūōku
  - As0014 20039, Iruma-gun
  - As0014 20036, Kawachi-Nagano
  - As0014 20045, Kita-gun
  - As0014 20065, Kitakyushu
  - As0014 20037, Osaka
  - As0014 20084, Saga
  - As0014 20048, Saitama
  - As0014 20031, Sapporo
  - As0014 20032, Suita
- As0014 40034, Amsterdam, Netherlands
- Poland (8):
  - As0014 40038, Elblag
  - As0014 40042, Krakow
  - As0014 40037, Lublin
  - As0014 40044, Poznan
  - As0014 40040, Torun
  - As0014 40041, Warsaw
  - As0014 40039, Wroclaw
  - As0014 40043, Wroclaw
- Spain (4):
  - As0014 40045, A Coruña
  - As0014 40046, Córdoba
  - As0014 40048, Santiago de Compostela
  - As0014 40049, Seville
- Turkey (Türkiye) (3):
  - As0014 40052, Ankara
  - As0014 40053, Ankara
  - As0014 40050, Istanbul
- United Kingdom (3):
  - As0014 40057, Edinburgh
  - As0014 40056, Leeds
  - As0014 40055, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Result] Brown MA, Rudwaleit M, van Gaalen FA, Haroon N, Gensler LS, Fleurinck C, Marten A, Massow U, de Peyrecave N, Vaux T, White K, Deodhar A, van der Horst-Bruinsma I. Low uveitis rates in patients with axial spondyloarthritis treated with bimekizumab: pooled results from phase 2b/3 trials. Ann Rheum Dis. 2024 Nov 14;83(12):1722-1730. doi: 10.1136/ard-2024-225933. PMID 38977276
- [Result] Ramiro S, Poddubnyy D, Mease PJ, Lopez-Medina C, Kim M, Massow U, Taieb V, Kragstrup TW, McGonagle D. Sustained resolution of enthesitis and peripheral arthritis over 104 weeks with bimekizumab in axial spondyloarthritis. RMD Open. 2025 Oct 22;11(4):e005969. doi: 10.1136/rmdopen-2025-005969. PMID 41125403
- [Derived] Marzo-Ortega H, Navarro-Compan V, Dubreuil M, Mease PJ, Magrey M, Rudwaleit M, D'Agostino MA, Gaffney K, Kay J, de la Loge C, Massow U, Taieb V, Vaux T, Deodhar A. Sustained improvements in spinal pain, morning stiffness, fatigue, sleep, physical function and overall health-related quality of life with bimekizumab in patients with axial spondyloarthritis: 2-year results from two phase 3 studies. RMD Open. 2025 Nov 28;11(4):e006013. doi: 10.1136/rmdopen-2025-006013. PMID 41314667
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794